CLINICAL TRIAL: NCT05153889
Title: Low Risk Non ST Elevation Myocardial Infarction With or Without Intensive Care Unit Admission : a Randomized Study
Brief Title: Low Risk Non ST Elevation Myocardial Infarction With or Without Intensive Care Unit Admission
Acronym: SELECTNSTEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0270; 2021-A02234-37 (Other: IDRCB)
Record Dates: First submitted 2021-10-27; First posted 2021-12-10 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-ST Elevated Myocardial Infarction
Keywords: Intensive Care Unit; General Cardiology Ward; ECG monitoring; Low risk NSTEMI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Hospitalization; Intensive Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive care unit (Other): systematic intensive care unit (ICU) monitoring
  Interventions: Other: Hospitalized in Intensive care unit
- General cardiology ward (Experimental): Group without ECG monitoring
  Interventions: Other: Hospitalized in General cardiology ward

INTERVENTIONS:
Other: Hospitalized in Intensive care unit — Patient hospitalized in Intensive care unit with ECG monitoring
  Arms: Intensive care unit
Other: Hospitalized in General cardiology ward — Patient hospitalized in General cardiology ward without ECG monitoring. patients randomized in this group will not be hospitalized in intensive care unit unless an event require intensive care unit monitoring.
  Arms: General cardiology ward

SUMMARY:
Favourable in-hospital outcome is observed in numerous patients after Non ST myocardial infarction (NSTEMI) with invasive strategy but European guidelines proposed systematic intensive care unit monitoring up to 24 h in lower risk patients (grade 1, level of evidence C). Regarding absence of prospective study supporting this strategy, we assessed the hypothesis that the lower risk NSTEMI patients identified through simple medical criteria and after coronary angiography evaluation may not require intensive care unit admission.

DETAILED DESCRIPTION:
The incidence of serious in hospital complications after NSTEMI has dramatically decreased over the past decades mainly due to early coronary angioplasty with new generation drug eluting stents surrounded by an optimal antithrombotic treatment (1). Major in-hospital adverse events after NSTEMI became uncommon and above all appears predictable including unstable hemodynamic state, acute stent thrombosis and life threatening arrhythmia (5-7). Recent 2020 European guidelines recommended that all patients with NSTEMI should be monitored up to 24 hours or up to percutaneous coronary intervention (PCI) in the intensive care unit (ICU) and rhythm monitoring > 24 h in patients at intermediate or high risk of cardiac arrhythmia (2). However, the usefulness of systematic ICU admission and ECG monitoring, for lower risk patients particularly when they have been stabilized with successful (PCI) has never been evaluated in a randomized study and remain controversial (8-10).

The main objective of this randomized study is to validate the feasibility and safety of a strategy without intensive care unit admission of lower risk NSTEMI patients after coronary angiography evaluation and successful PCI when required, compared to the conventional strategy using systematic ICU monitoring.

All patients admitted in our hospital for NSTEMI (initial admission of patients in ICU or directly in the cath lab) will have systematic coronary angiography evaluation and PCI when required. They will be classified as low or high risk patients related to guidelines derived criteria including results of coronary angiography evaluation. Low risk patients will be randomized in ICU admission group (control group) or general cardiology ward (GCW) group (experimental group) without ECG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18 years
* NSTEMI was defined according guidelines with chest pain with or without ECG modifications and significant troponin elevation (hs-cTn T *≥ 52 ng/l) or significant variation > 10 ng/l between 2 dosages between 1 or 3 hours interval) * Elecsys Roche
* Coronary angiography mandatory < 24 h after first troponin assay according to 2020 NSTEMI guidelines and PCI if required
* Low risk NSTEMI defined with (all necessary):

  * Age<85 years
  * Optimal antithrombotic therapy using new generation P2Y12 inhibitors (ticagrelor or prasugrel) or clopidogrel and aspirin with preloading at the latest before PCI
  * Success of PCI (one or 2 arteries)
  * Low risk of severe arrhythmia (ESC criteria) if none of the following criteria: haemodynamically unstable, major arrhythmias, LVEF <40%, failed reperfusion, additional critical coronary stenosis of major vessels, complications related to percutaneous revascularization,
  * No major comorbidities requiring specific care
  * Success of PCI without any event within 30 minutes after the procedure
  * Low bleeding risk (ESC criteria) according to CRUSADE criteria validated in NSTEMI

Exclusion Criteria:

* STEMI
* Unstable angina troponin <5ng/l* or <14ng/l with variation <4ng/l between 2 dosages )* Elecsys Roche
* High risk NSTEMI if one low risk criteria defined above is absent
* Patient with acute coronary syndromes (ACS) requiring transfer to resuscitation unit and not to intensive care unit for any reason
* Coronary angiography not performed or performed > 24 h after first troponin assay in ICU
* Pregnant or breastfeeding woman
* Patient unable or refusing to sign inform consent
* Patient without health care insurance
* Patient under legal guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Success of the experimental strategy defined by absence of major adverse events 4 +/- 3 days after inclusion | 4 +/- 3 days after inclusion
  Major adverse events include : mortality (total and cardiovascular), severe bleeding (BARC criteria >2), major vascular events (BARC 3 or 4 criteria) , cardiac failure requiring specific therapy ,acute kidney injury (RAKIN classification ≥grade 2) , major neurologic events confirmed with brain imaging, severe conductive or rhythm disorder, new coronary ischemic event requiring coronary angiography, any medical decision for secondary ICU transfer

SECONDARY OUTCOMES:
Incidence of low vs high risk NSTEMI patients admitted in ICU or in cath lab | 1 month follow up
  number of low vs high risk NSTEMI (flow chart)
Incidence of each event included in the combined primary outcome | 1 month follow up
  evaluation of each event of combined primary end point
Comparison of hospitalization length of stay for the 2 groups | though hospital follow up, an average of 5 days
  lenght of stay in ICU and total hospitalization stay in days
ICU length of stay in the control group | though hospital follow up, an average of 5 days
  ICU length of stay in the control group in days
Evolution of patient satisfaction (questionnaire) | 1 month +/- 7 days after inclusion
  a short 5 questions by phone regarding satisfaction in the 2 groups
Comparison of total mortality in both arm | 1 month +/- 7 days after inclusion
  total mortality in both arms
Comparison of cardiovascular mortality in both arm | 1 month +/- 7 days after inclusion
  cardiovascular mortality in both arms
Comparison of new hospitalization for cardiac event in both arms | 1 month +/- 7 days after inclusion
  new hospitalization for cardiac reasons
Comparison of direct medical cost of the initial inpatient stay in both arm | during hospitalization stay
  economic study regarding medical cost

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - UH Nîmes, Nîmes, Gard
  - UH Montpellier, Montpellier
  - UH Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harvey S, Harrison DA, Singer M, Ashcroft J, Jones CM, Elbourne D, Brampton W, Williams D, Young D, Rowan K; PAC-Man study collaboration. Assessment of the clinical effectiveness of pulmonary artery catheters in management of patients in intensive care (PAC-Man): a randomised controlled trial. Lancet. 2005 Aug 6-12;366(9484):472-7. doi: 10.1016/S0140-6736(05)67061-4. PMID 16084255
- [Background] Bonnefoy-Cudraz E, Bueno H, Casella G, De Maria E, Fitzsimons D, Halvorsen S, Hassager C, Iakobishvili Z, Magdy A, Marandi T, Mimoso J, Parkhomenko A, Price S, Rokyta R, Roubille F, Serpytis P, Shimony A, Stepinska J, Tint D, Trendafilova E, Tubaro M, Vrints C, Walker D, Zahger D, Zima E, Zukermann R, Lettino M. Editor's Choice - Acute Cardiovascular Care Association Position Paper on Intensive Cardiovascular Care Units: An update on their definition, structure, organisation and function. Eur Heart J Acute Cardiovasc Care. 2018 Feb;7(1):80-95. doi: 10.1177/2048872617724269. Epub 2017 Aug 17. PMID 28816063
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058